CLINICAL TRIAL: NCT04880031
Title: A Phase 2a, Randomized, Blinded, Placebo-controlled Study of BOS-580 in Obese Subjects at Risk for, or With Biopsy-confirmed, Nonalcoholic Steatohepatitis (NASH) With a Single Arm Open-label Extension
Brief Title: A Study of BOS-580 in Obese Subjects at Risk for, or With Biopsy-confirmed, Nonalcoholic Steatohepatitis (NASH) With an Extension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boston Pharmaceuticals (Industry)
Collaborators: GSK Research and Development Limited (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 301182 (BOS-580-201)
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
Keywords: BOS-580; Safety; Tolerability; Pharmacokinetics; Efimosfermin
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Part C - Open Label; Part D - Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort A1: Efimosfermin Dose 1 or placebo (PBO) (Experimental)
  Interventions: Drug: Efimosfermin; Drug: Placebo
- Cohort A2: Efimosfermin Dose 2 or PBO (Experimental)
  Interventions: Drug: Efimosfermin; Drug: Placebo
- Cohort A3: Efimosfermin Dose 3 or PBO (Experimental)
  Interventions: Drug: Efimosfermin; Drug: Placebo
- Cohort A4: Efimosfermin Dose 4 or PBO (Experimental)
  Interventions: Drug: Efimosfermin; Drug: Placebo
- Cohort A5: Efimosfermin Dose 5 or PBO (Experimental)
  Interventions: Drug: Efimosfermin; Drug: Placebo
- Part B: Efimosfermin Dose 1 or PBO (Experimental)
  Interventions: Drug: Efimosfermin; Drug: Placebo
- Part C: Efimosfermin Dose 1 (Experimental)
  Interventions: Drug: Efimosfermin
- Part D: Efimosfermin Dose 6 or PBO (Experimental)
  Interventions: Drug: Efimosfermin; Drug: Placebo
- Part D: Efimosfermin Dose 1 or PBO (Experimental)
  Interventions: Drug: Efimosfermin; Drug: Placebo

INTERVENTIONS:
Drug: Efimosfermin — Efimosfermin will be administered by subcutaneous injection
  Other Names: BOS-580
Drug: Placebo — Placebo will be administered by subcutaneous injection
  Arms: Cohort A1: Efimosfermin Dose 1 or placebo (PBO); Cohort A2: Efimosfermin Dose 2 or PBO; Cohort A3: Efimosfermin Dose 3 or PBO; Cohort A4: Efimosfermin Dose 4 or PBO; Cohort A5: Efimosfermin Dose 5 or PBO; Part B: Efimosfermin Dose 1 or PBO; Part D: Efimosfermin Dose 1 or PBO; Part D: Efimosfermin Dose 6 or PBO

SUMMARY:
This is a randomized, blinded, placebo-controlled study of Efimosfermin in obese participants at risk for, or with biopsy-confirmed, nonalcoholic steatohepatitis (NASH), with a single arm open-label extension. It includes Parts A, B, C and D.

ELIGIBILITY:
Inclusion Criteria (Part A and Part B):

* Participant is either male or female and 18 to 75 years of age inclusive, at the time of signing the informed consent
* Obese participants with body mass index (BMI) of ≥ 27 kg/m^2
* Hepatic fat fraction (HFF) measured by magnetic resonance imaging derived proton density fat fraction (MRI-PDFF) ≥8%
* Liver fibrosis assessment based on a vibration controlled transient elastography (VCTE) liver stiffness measurement (LSM) score of 7.0 to 9.9 kPa (Part A only) inclusive or 7.0 to 20.0 kPa (Part B only) inclusive and Liver injury assessment measured by aspartate aminotransferase (AST) >25U/L. A qualifying historical biopsy (confirmed eligibility based on the central pathology read) supersedes the LSM, controlled attenuation parameter (CAP) score criteria and AST criteria.
* Histopathologically confirmed F2 or F3 stage NASH on a diagnostic liver biopsy performed during Screening or within 6 months prior to the first day of dosing for historical biopsies (Part B only).
* History or presence of at least 2 of 4 components of metabolic syndrome: obesity/overweight, dyslipidemia (high triglycerides and/or low high density lipoprotein [HDL]), type 2 diabetes with elevated glycated hemoglobin (HbA1c), and hypertension.

Inclusion Criteria (Part C):

* Participant must have completed the Part B of the study.
* Participant willing to undergo liver biopsy at Week 56
* NASH F stage <F4 at 24 week assessment in Part B

Inclusion Criteria (Part D):

* BMI of ≥ 25 kg/m^2
* Liver fibrosis based on assessments taken during screening visit
* Participant should be willing and able to undergo liver biopsy during Screening (if a historical biopsy within 12 months prior to Screening is not available) and per protocol as judged by the Investigator.
* Other inclusion criteria may apply

Exclusion Criteria (Part A and Part B):

* Documented clinical, laboratory or radiologic evidence of cirrhosis (compensated or decompensated)
* Triglycerides ≥ 500 mg/dL
* Change in body weight (more than 5% self-reported OR 5 kg self-reported change during the previous 3 months from Screening, whichever is smaller)
* History of type 1 diabetes, diabetic ketoacidosis, or positive glutamic acid decarboxylase (GAD) auto-antibodies (latent autoimmune diabetes in adults)
* Hemoglobin A1c > 9.5%
* Participants with a condition that requires substantial anticoagulant medication may not be eligible for the study enrollment (e.g., deep vein thrombosis).

Exclusion Criteria (Part C):

• Participants that received their 24 week dose in Part B > 10 weeks prior to enrollment into Part C

Exclusion Criteria (Part D):

* Other causes of chronic liver disease
* Documented evidence or history of decompensated liver cirrhosis.
* History of type 1 diabetes or poorly controlled type 2 diabetes.
* History of malignancy.
* Use of other investigational drugs.
* Other exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2025-10-27 (Actual)

PRIMARY OUTCOMES:
Part A, Part B, Part C, and Part D: Number of participants with treatment-emergent adverse events (TEAEs) and treatment-emergent serious adverse events (TESAEs) | Until End of study/Early Termination (Day 393)
  The effects of Efimosfermin on safety and tolerability will be assessed.
Part A, Part B, Part C, and Part D: Changes from Baseline in systolic and diastolic blood pressure (BP) | Baseline, Week 12 (Day 85, Part A), Week 24 (Day 169, Part B), Week 56 (Day 393, Part C), and Weeks 36 (Day 253), and 48 (Day 337) (Part D)
  The effects of Efimosfermin on safety and tolerability will be assessed.
Part A, Part B, Part C, and Part D: Changes from Baseline in heart rate | Baseline, Week 12 (Day 85, Part A), Week 24 (Day 169, Part B), Week 56 (Day 393, Part C), and Weeks 36 (Day 253), and 48 (Day 337) (Part D)
  The effects of Efimosfermin on safety and tolerability will be assessed.
Part A, Part B, Part C, and Part D: Number of participants with Grade 3 and Grade 4 laboratory abnormalities | Baseline, Week 12 (Day 85, Part A), Week 24 (Day 169, Part B), Week 56 (Day 393, Part C), and Weeks 36 (Day 253), and 48 (Day 337) (Part D)
  The effects of Efimosfermin on safety and tolerability will be assessed.

SECONDARY OUTCOMES:
Part A only: Efimosfermin serum concentration on Day 8 of the first dose | Day 8
  The pharmacokinetics (PK) of Efimosfermin will be assessed.
Part A only: Efimosfermin serum concentration at the end of the dosing interval (Ctrough) | Pre-dose at Days 15, 29, 43, 57, 71, 85 and 113 (End of study/Early termination) for bi-weekly schedule; pre-dose on Days 29, 57, 85 and 113 (End of study/Early termination) for the monthly schedule
  The PK of Efimosfermin will be assessed.
Part B only: Efimosfermin serum concentration on Day 7 | Day 7
  The PK of Efimosfermin will be assessed.
Part B and Part C: Efimosfermin serum concentration at the end of the dosing interval (Ctrough) | Pre-dose at Days 29, 57, 85, 113, 141, 169, 225, 253, 281, 309, 316, 323, 330, 337, 365 and at Day 393 (End of study/Early Termination)
  The PK of Efimosfermin will be assessed.
Part B and Part C: Area under the serum concentration-time curve (AUC) for Efimosfermin for one dosing interval at steady state | At Days 121, 127, 134, 316, 323, 330 and pre-dose at Days 141 and 337
  The PK of Efimosfermin will be assessed.

CONTACTS AND LOCATIONS:
Locations (48):
- United States (48):
  - Central Research Associates, Birmingham, Alabama
  - Arizona Liver Health, Chandler, Arizona
  - Arizona Liver Health, Peoria, Arizona
  - Arizona Liver Health, Tucson, Arizona
  - Liver Institute PPLC, Tucson, Arizona
  - QLMC, Tucson, Arizona
  - Alliance Research Institute, Canoga Park, California
  - Ark Clinical Research, Fountain Valley, California
  - Fresno Clinical Research Center, Fresno, California
  - Catalina Research Institute, Montclair, California
  - Knowledge Research Center, Orange, California
  - FOMAT Medical Research, Oxnard, California
  - Inland Empire Clinical Trials, Rialto, California
  - Southwest General Healthcare Center, Fort Myers, Florida
  - Covenant Metabolic Specialists - Fort Myers, Fort Myers, Florida
  - Evolution Clinical Trials, Hialeah Gardens, Florida
  - Entrust Clinical Research Center, Kendall, Florida
  - Galenus Group, Lehigh Acres, Florida
  - G+C Research Group, Miami, Florida
  - Miami Clinical Research, Miami, Florida
  - Advanced Clinical Research, Miami, Florida
  - Admed Research, Miami, Florida
  - Century Research, Miami, Florida
  - Panex Clinical Research, Miami Lakes, Florida
  - Charter Research, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Covenant Metabolic Specialists - Sarasota, Sarasota, Florida
  - Tandem Clinical Research, Marrero, Louisiana
  - Kansas City Research Institute, Kansas City, Missouri
  - Coastal Research Institute, LLC, Fayetteville, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Velocity Clinical Research, East Greenwich, Rhode Island
  - Accelemed Research, Austin, Texas
  - Pinnacle Clinical Research - Austin, Austin, Texas
  - Texas Liver Institute - Austin, Austin, Texas
  - Apex Mobile Clinical Research, Bellaire, Texas
  - South Texas Research Institute-Brownsville, Brownsville, Texas
  - South Texas Research Institute-Edinburg, Edinburg, Texas
  - Pinnacle Clinical Research - Georgetown, Georgetown, Texas
  - Houston Research Institute, Houston, Texas
  - LinQ Research, LLC, Pearland, Texas
  - Quality Research, Inc, San Antonio, Texas
  - American Research Corporation at Texas Liver Institute, San Antonio, Texas
  - Pinnacle Clinical Research - San Antonio, San Antonio, Texas
  - Velocity Clinical Research - Waco, Waco, Texas
  - Olympus Family Medicine, Salt Lake City, Utah
  - South Ogden Family Medicine, South Ogden, Utah
  - Liver Institute NorthWest, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Noureddin M, Kowdley KV, Odrljin T, Bain G, Zhao J, Jeglinski B, Koziel MJ, Loomba R. Efimosfermin alfa (BOS-580) once per month in people with metabolic dysfunction-associated steatohepatitis with F2 or F3 fibrosis: results from a 24-week, randomised, double-blind, placebo-controlled, phase 2 trial. Lancet. 2026 Feb 5:S0140-6736(25)02276-7. doi: 10.1016/S0140-6736(25)02276-7. Online ahead of print. PMID 41655584
- [Derived] Loomba R, Kowdley KV, Rodriguez J, Kim NJ, Alvarez AM, Morrow L, Jeglinski B, Clawson A, Chowdhury S, Bain G, Odrljin T. Efimosfermin alfa (BOS-580), a long-acting FGF21 analogue, in participants with phenotypic metabolic dysfunction-associated steatohepatitis: a multicentre, randomised, double-blind, placebo-controlled, phase 2a trial. Lancet Gastroenterol Hepatol. 2025 Aug;10(8):734-745. doi: 10.1016/S2468-1253(25)00067-6. Epub 2025 Jun 6. PMID 40484014